CLINICAL TRIAL: NCT01903330
Title: A Randomized, Double-blinded, Placebo-controlled Study of (ERC1671/GM-CSF/Cyclophosphamide)+Bevacizumab vs. (Placebo Injection/Placebo Pill) +Bevacizumab in the Treatment of Recurrent/Progressive, Bevacizumab naïve Glioblastoma Multiforme and Glioasarcoma Patients (WHO Grade IV Malignant Gliomas, GBM)
Brief Title: ERC1671/GM-CSF/Cyclophosphamide for the Treatment of Glioblastoma Multiforme
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Epitopoietic Research Corporation (Industry)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCI13-14 ERC1671-H02 2013-9863; UCI 13-14 (Other: University of California, Irvine); 2013-9863 (Other: University of California, Irvine)
Record Dates: First submitted 2013-06-26; First posted 2013-07-19 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: ERC1671; GM-CSF; Cyclophosphamide; Bevacizumab
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Cyclophosphamide; Sucrose; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (ERC1671/GM-CSF/Cyclophosphamide)+bevacizumab/bevacizumab biosimilar (Experimental): ERC1671 and GM-CSF will be intradermally administered, while cyclophosphamide is orally administered. GM-CSF dose is 500mcg fixed dose and cyclophosphamide dose is 50 mg/day. Bevacizumab or approved bevacizumab biosimilars are administered as standard of care at 10 mg/kg every 2 weeks.
  The treatment will be repeated every 28 days until progression of disease or intolerance.
  Interventions: Drug: ERC1671; Drug: GM-CSF; Drug: Cyclophosphamide; Drug: Bevacizumab/Bevacizumab Biosimilar
- (Placebo Injection/Placebo Pill) +Bevacizumab/bevacizumab biosimilar (Placebo Comparator): The control group will have the same study schedule except that the patients will be receiving the Oral Control on the Cyclophosphamide treatment days and the Injectable control on the GM-CSF + ERC1671 treatment days. The control group will receive bevacizumab or approved bevacizumab biosimilar just as the active treatment group above.
  The treatment will be repeated every 28 days until progression of disease or intolerance.
  Interventions: Drug: Oral Control (Sucrose pill); Drug: Injectable control (Sodium Chloride Injection United States Pharmacopeia (USP) (0.9%)); Drug: Bevacizumab/Bevacizumab Biosimilar

INTERVENTIONS:
Drug: ERC1671 — Given intradermally
  Other Names: Gliovac
  Arms: (ERC1671/GM-CSF/Cyclophosphamide)+bevacizumab/bevacizumab biosimilar
Drug: GM-CSF — Given intradermally
  Other Names: Leukine®; sargramostim
  Arms: (ERC1671/GM-CSF/Cyclophosphamide)+bevacizumab/bevacizumab biosimilar
Drug: Cyclophosphamide — Given PO. Drug class: Alkylating Agent; Antineoplastic Agent; Nitrogen Mustard.
  Other Names: 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Arms: (ERC1671/GM-CSF/Cyclophosphamide)+bevacizumab/bevacizumab biosimilar
Drug: Oral Control (Sucrose pill) — Given PO
  Arms: (Placebo Injection/Placebo Pill) +Bevacizumab/bevacizumab biosimilar
Drug: Injectable control (Sodium Chloride Injection United States Pharmacopeia (USP) (0.9%)) — Given IV
  Arms: (Placebo Injection/Placebo Pill) +Bevacizumab/bevacizumab biosimilar
Drug: Bevacizumab/Bevacizumab Biosimilar — Given IV. Drug class: Immunological Agent; Monoclonal Antibody.
  Other Names: Avastin; MVASI; bevacizumab-awwb; bevacizumab-bvzr; ZIRABEV

SUMMARY:
This phase II clinical trial studies how well ERC1671 plus Granulocyte-macrophage colony-stimulating factor (GM-CSF) plus Cyclophosphamide with Bevacizumab works compared to Placebo Injection plus Placebo Pill with Bevacizumab in treating patients with recurrent/progressive, bevacizumab naïve glioblastoma multiforme and gliosarcoma (World Health Organization (WHO) grade IV malignant gliomas, GBM).

DETAILED DESCRIPTION:
This is a blinded Phase II study of ERC1671 in combination with bevacizumab in patients with relapsed, bevacizumab naive glioblastoma. The patients who will be randomized (in a 1:1 ratio) to receive either ERC 1671 in combination with GM-CSF and cyclophosphamide or a placebo control, in combination with bevacizumab. The study will be double blinded.

ERC1671/GM-CSF will be intradermally administered, while cyclophosphamide is orally administered. GM-CSF dose is 500mcg fixed dose and cyclophosphamide dose is 50 mg/day. Bevacizumab or approved bevacizumab biosimilars are administered as standard of care at 10 mg/kg every 2 weeks.

The treatment cycles will be 28 days long.

ELIGIBILITY:
Inclusion Criteria:

-Patients must have histologically confirmed diagnosis of a recurrent/progressive WHO grade IV malignant gliomas (glioblastoma multiforme and gliosarcoma) and meet the following inclusion criteria:

1. Age ≥18 years of age.
2. Histologic diagnosis of glioblastoma or gliosarcoma (WHO Grade IV).
3. KPS of ≥ 70%.
4. Life expectancy > 12 weeks.
5. First or second relapse of glioblastoma.
6. Previous treatment for glioblastoma must include surgery (biopsy, partial resection, or full surgical resection), conventional radiation therapy and temozolomide (TMZ).
7. MRI record must be obtained showing the MRI was conducted at least 4 weeks after any salvage surgery, and at least 12 weeks after radiation therapy, or at least 4 weeks after radiation for a new lesion outside the prior primary radiation field unless relapse is confirmed by tumor biopsy or new lesion outside of radiation field, or if there are two MRIs confirming progressive disease per iRANO that are 8 weeks apart
8. If prior therapy with gamma knife or other focal high-dose radiation, must have subsequent histologic documentation of local relapse, or relapse with new lesion outside the irradiated field.
9. Resolution of all chemotherapy or radiation-related toxicities ≤ CTCAE Grade 1 severity, except for alopecia and hematologic toxicity. Patients taking temozolomide can start study treatment 23 days from the last temozolamide dose.For all other chemotherapy drugs, study treatment can start as long as all adverse events related to their prior treatment are no higher than Grade 1.
10. Systemic corticosteroid therapy must be at a dose of ≤ 4 mg of dexamethasone or equivalent per day during the week prior to Day 1.
11. Pre-surgical Bi-dimensionally measurable disease (as per iRANO criteria)
12. Patients must have normal organ and marrow function as defined below:

    * hemoglobin (Hbg) > 9g/dL,
    * leukocytes >1,500/mcL
    * absolute neutrophil count>1,000/mcL
    * CD4 count > 450/mcL
    * platelets>125,000/mcL
    * Serum bilirubin = 1.5 × upper limit of normal (ULN) or = 3 x ULN if Gilbert's disease is documented AST(SGOT) and ALT(SGPT)<2.5 X institutional upper limit of normal
    * serum creatinine < 1.5 mg/dl
13. Signed informed consent approved by the Institutional Review Board;
14. If sexually active, patients must agree to take contraceptive measures for the duration of the treatments.

Exclusion Criteria:

1. Subjects unable to undergo an MRI with contrast.
2. Presence of diffuse leptomeningeal disease
3. History, presence, or suspicion of metastatic disease
4. Administration of immunosuppressive drugs less than 2 weeks prior to first dose of ERC1671, except dexamethasone for cerebral edema as detailed above;
5. Prior receipt of bevacizumab, or bevacizumab biosimilars or other VEGF- or VEGF receptor-targeted agents
6. Known contraindication or hypersensitivity to any component of bevacizumab.
7. Evidence of recent hemorrhage on screening MRI of the brain with the following exceptions: presence of hemosiderin; resolving hemorrhagic changes related to surgery; presence of punctate hemorrhage in the tumor.
8. Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1.
9. Evidence of bleeding diathesis or coagulopathy as documented by an elevated PT, PTT or bleeding time and clinically significant;
10. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1.
11. Urine protein: creatinine ratio ≥ 1.0 at screening;
12. Anticipation of need for major surgical procedure during the course of the study.
13. Serious non-healing wound, ulcer, or bone fracture.
14. Active infection requiring treatment, known immunosuppressive disease, active systemic autoimmune diseases such as lupus, receipt of systemic immunosuppressive therapy, human immunodeficiency virus (HIV) infection, Hepatitis B or Hepatitis C
15. Uncontrolled hypertension, blood pressure of > 150 mmHg systolic and > 100 mmHg diastolic, or history of hypertensive encephalopathy. Subjects with any known uncontrolled inter-current illness including ongoing or active infection, symptomatic congestive heart failure (NYHA Gr.2 or >), myocardial infarction, unstable angina pectoris , within the past 12 months
16. Stroke, transient ischemic attack, unstable angina, myocardial infarction or congestive heart failure (New York Heart Association Grade II or greater) within the past 6 months.Unstable or severe intercurrent medical conditions chronic renal disease, or uncontrolled diabetes mellitus.
17. Women who are pregnant or lactating. All female patients with reproductive potential must have a negative pregnancy test prior to Day 1 and must use a reliable form of contraception during study participation.
18. Men refusing to exercise a reliable form of contraception.
19. History of any malignancy (other than glioblastoma) during the last three years except non-melanoma skin cancer, in situ cervical cancer, treated superficial bladder cancer or cured, early-stage prostate cancer in a patient with Prostate Surface Antigen (PSA) level <ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-03; Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival at 12 months of patients with recurrent, bevacizumab naïve glioblastoma treated with ERC1671 in combination with GM-CSF and cyclophosphamide plus bevacizumab as compared with patients receiving bevacizumab plus placebo controls. | 12 months
  To evaluate overall survival in patients with with recurrent, bevacizumab naïve glioblastoma treated with ERC1671 in combination with GM-CSF and cyclophosphamide plus bevacizumab as compared with patients receiving bevacizumab plus placebo controls.

SECONDARY OUTCOMES:
Rate of Progression-Free Survival | 12 months
  Progression-free survival will be defined as the time from Day 1 to the date of progression or death due to any cause.
Immune Response | 12 months
  The patient's immune response evaluation will include cytotoxic T lymphocytes (CTL) (CD3+/cluster of differentiation (CD)8+) and Treg (CD3+/CD4+/cluster of differentiation 25+ (CD25+)/CD127low) populations where CD refers to cluster of differentiation. Cytokine analyses should initially be limited to IFN-ɣ, TNF and IL-6. Further immune studies should include transforming growth factor (TGF)-B2, IL-12, IL-10.
Percentage of Grade 3-5 Adverse Events | 12 months
  Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0. Safety will also be assessed by clinical laboratory tests, physical examinations, vital sign measurements and the incidence and severity of adverse events (AEs).
Rate of Radiographic Response as assessed using MacDonald Criteria or IRANO | 12 month
  Patients will be followed both clinically and radiographically every 6 weeks for evidence of tumor progression. Tumor response will be assessed using the MacDonald Criteria or iRANO, Immunotherapy Response Assessment in Neuro-Oncology.
  iRANO/MacDonald CRITERIA:
  * Complete response (CR): Disappearance of all enhancing tumor on contrast enhanced MRI scan.
  * Partial response (PR): Greater than or equal to a 50% reduction in the size (sum of products of the largest diameter, SPD) for all enhancing lesions.
  * Stable Disease (SD): SPD <50% decrease to <25% increase, does not qualify for CR, PR, or progression.
  * Progressive Disease (PD): Greater than or equal to a 25% increase in SPD.
  * Unable to Assess (UA): Some target lesions cannot be evaluated because of technical factors.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela A. Bota, MD, PhD, Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - University of California, Irvine, Orange, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schijns VE, Pretto C, Devillers L, Pierre D, Hofman FM, Chen TC, Mespouille P, Hantos P, Glorieux P, Bota DA, Stathopoulos A. First clinical results of a personalized immunotherapeutic vaccine against recurrent, incompletely resected, treatment-resistant glioblastoma multiforme (GBM) tumors, based on combined allo- and auto-immune tumor reactivity. Vaccine. 2015 May 28;33(23):2690-6. doi: 10.1016/j.vaccine.2015.03.095. Epub 2015 Apr 10. PMID 25865468